CLINICAL TRIAL: NCT06841237
Title: Randomized Controlled Trial on the Efficacy and Safety of Xiang Lei Ointment in Diabetic-related Ulcer Management
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Long Zhang, Professor, Head of Wound Healing Center, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Long2025-DRW-xianglei
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Diabetic Wound; Wound Infection; Wound Heal
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Experimental): Clinical standard treatment protocols plus Xiang Lei Ointment
  Interventions: Other: Xiang Lei Ointment plus Clinical standard treatment protocols
- control group (Sham Comparator): Clinical standard treatment protocols
  Interventions: Other: Clinical standard treatment protocols

INTERVENTIONS:
Other: Xiang Lei Ointment plus Clinical standard treatment protocols — A therapy for chronic wound healing
  Arms: test group
Other: Clinical standard treatment protocols — A therapy for chronic wound healing
  Arms: control group

SUMMARY:
Diabetes is one of the major chronic diseases. Diabetic ulcers are important adverse outcomes of diabetes. Approximately 80% of lower - limb amputations are caused by diabetic foot ulcers, which are the main causes of disability and death among patients. Moreover, it places a huge burden on the medical insurance system. Currently, there are western medicine treatment guidelines for diabetic foot, yet the clinical efficacy is less than satisfactory. The amputation rate caused by diabetic foot ulcers continues to rise every year. There is an urgent clinical need for novel and effective intervention measures to address this disease.

Macrophages are important cells involved in the inflammatory and proliferative phases of wounds, playing a crucial role in wound repair and reconstruction. Diabetes can cause wounds to remain in the pro - inflammatory stage continuously, leading to the aggregation of M1 macrophages and preventing their timely transformation into the pro - proliferative and repair stage. As a result, wounds exhibit persistent chronic inflammation and delayed tissue proliferation or remodeling.

Xianglei Tangzu Ointment is a natural medicine approved for marketing by the National Medical Products Administration in November 2023. Its ingredients include Pogostemon cablin extract and asiaticoside. Research shows that the plant components in Xianglei Tangzu Ointment can promote the transformation of M1 macrophages into M2 macrophages, thereby reducing the inflammatory response and accelerating the proliferative repair of diabetic wounds. It has achieved certain curative effects in the clinical treatment of promoting wound healing. In order to use Xianglei Tangzu Ointment more precisely, accumulate clinical evidence - based medicine evidence, and explore the effectiveness and safety of Xianglei Tangzu Ointment in treating diabetic ulcers under the guidance of the chronic wound staging theory, clinical evidence - based medicine evidence needs to be obtained.

ELIGIBILITY:
Inclusion Criteria:

* a confirmed diagnosis of type 1 or type 2 diabetes mellitus that meets the standard World Health Organization definition, with blood glucose controlled prior to enrolment and a glycated haemoglobin HbA1c level of less than 10%;
* the type of wound is an ulcer;
* the wound etiology is diabetic, mainly abnormalities in blood glucose, resulting in poor or prolonged healing and requiring standard wound therapy;
* the staging of the wound is in the granulation phase;
* voluntary participation in the study and signing of an informed consent form.

Exclusion Criteria:

* acute heart attack, heart failure, hepatitis, shock, expiratory failure and other serious diseases that have not been corrected;
* uncontrolled blood glucose, fasting blood glucose > 15 mmol/L and glycated haemoglobin > 12%;
* active bleeding in the wound, which does not allow the implementation of the conventional basic treatment plan;
* serum albumin < 20 g/L; haemoglobin < 60 g/L; platelets < 50 x 109/L;
* a state of disseminated infection that is being or will be treated with antibiotics
* patients with advanced malignant tumours;
* active autoimmune disease;
* previous allergy to topical human granulocyte macrophage stimulating factor gel (Jinfuning);
* inability of the patient to co-operate or mental disorder;
* in the judgement of the investigator, the subject has a clearly irremovable cause of wound healing, is unsuitable for the study or is unable to comply with the requirements of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
wound area reduction rate | From enrollment to the end of treatment at 2 weeks
  Pre-treatment area minus post-treatment area, then divided by pre-treatment area

SECONDARY OUTCOMES:
wound healing rate | From enrollment to the end of treatment at 3 weeks
  Percentage of healed wounds to total cases by D21
Granulation tissue status | From enrollment to the end of treatment at 3 weeks
  They were classified as healthy granulation, inflammatory granulation, infected granulation, oedematous granulation, and aged granulation. D0/D14/D21, wound granulation tissue status was recorded separately
wound infection control | From enrollment to the end of treatment at 3 weeks
  0 points for no infection, 1 point for reduction of localised infection; 2 points for maintenance or exacerbation of localised infection; 3 points for disseminated infection; record D0/D14/D21, the status of the wound infection and record the scoring results respectively

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University 3rd Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No